CLINICAL TRIAL: NCT05416580
Title: Randomized, Double-blind, Placebo-controlled Study of Ursodeoxycholic Acid (UDCA) Therapy on Biomarkers of Oxidative Stress, Inflammatory and Endothelial Dysfunction in Patients With Type 2 Diabetes Mellitus
Brief Title: Efficacy of Ursodeoxycholic Acid (UDCA) in Patients With Type 2 Diabetes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Banja Luka (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UDCA01T2DM
Record Dates: First submitted 2022-05-30; First posted 2022-06-13 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2022-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; UDCA; Metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Ursodeoxycholic Acid; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UDCA + metformin (Experimental): UDCA in addition to Metformin Treatment
  All subjects will be treated with UDCA 1500 mg/day, and Metformin, up to 2000 mg/day, by oral administration, respectively, for 8 weeks.
  Interventions: Drug: UDCA (Ursodeoxycholic acid); Drug: Metformin
- Placebo + metformin (Placebo Comparator): Placebo of UDCA in addition to Metformin Treatment
  All subjects will be treated with a Placebo of UDCA, and Metformin, up to 2000 mg/day, by oral administration, respectively, for 8 weeks.
  Interventions: Drug: Placebo; Drug: Metformin

INTERVENTIONS:
Drug: UDCA (Ursodeoxycholic acid) — UDCA is administered orally in addition to metformin therapy in the recommended doses in patients with type 2 diabetes mellitus.
  Other Names: Ursofalk; Bilexin
  Arms: UDCA + metformin
Drug: Placebo — Placebo is administered orally in addition to metformin therapy in the recommended doses in patients with type 2 diabetes mellitus.
  Arms: Placebo + metformin
Drug: Metformin — Metformin therapy is administered in the recommended dose in patients with type 2 diabetes mellitus.
  Other Names: Siofor; Glucophage

SUMMARY:
The purpose of this study is to evaluate the effects of ursodeoxycholic acid (UDCA) compared to placebo on biomarkers of oxidative stress, inflammation, and endothelial dysfunction in patients with type 2 diabetes mellitus (T2DM) who are treated with metformin but did not meet the target HbA1C < 7%.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double-blind, placebo-controlled, evaluation of the efficacy of UDCA on oxidative stress, inflammation, and endothelial dysfunction in combination with metformin after 8 weeks in patients with T2DM who did not meet HbA1C < 7%.

Study site: a single study center (Primary Health Care Institution in Banja Luka, as recruiter center) including Center for Biomedical Research, Faculty of Medicine University of Banja Luka, as reference coordinator and research center.

Sample size :

60 patients, randomized in a 1:1 allocation ratio.

Objectives

1. To investigate the effects of UDCA added to metformin on glycemia, HbA1C, Homeostatic Model Assessment for Insulin Resistance (HOMA-IR), lipoproteins, and body mass index.
2. To investigate whether UDCA has an impact on lipid peroxidation index, nitric oxide metabolites, hydrogen peroxide (H2O2), superoxide anion radical (O2-), and total antioxidant capacity.
3. To investigate whether UDCA has an impact on the dynamic of inflammatory markers interleukin-6 (IL-6), tumor necrosis factor-α (TNF-α), and high sensitive CRP (hsCRP).
4. To investigate whether UDCA has an impact on von Willebrand factor (vWF), Intercellular Adhesion Molecule 1 (ICAM-1), Vascular Adhesion Molecule 1 (VCAM-1), fibrinogen, homocysteine, folic acid, and vitamin D levels.

Treatments arms:

UDCA (1500 mg/day) + Metformin (maximum tolerated daily dose) UDCA placebo + Metformin (maximum tolerated daily dose)

Treatment duration :

8 weeks

Assessment - clinical and laboratory sampling:

Informed consent and Screening - 7 days prior to randomization

Study visits (V):

V1 - Randomization and Enrollment (Baseline) V2 - 4 weeks after Baseline V3 - 8 weeks after Baseline.

No interim analysis is planned. The analysis will be performed at the end of the study after data review and freezing of the database according to the intent to treat principle.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Type 2 Diabetes mellitus verified at least 1 year prior to the study enrollment
* Treatment with metformin at a maximally tolerated dose (up to 2000 mg/day) in patients with an incomplete biochemical response showing HbA1c ≥ 6,5%.
* Body mass index (BMI) corresponding to overweight and obesity (≥ 25 kg/m2)

Exclusion Criteria:

* Insulin treatment within 12 weeks prior to the study enrollment
* Treatment with Glucagon-like peptide 1 (GLP-1) analogs within 12 weeks prior to the study enrollment
* Systemic administration of glucocorticoids continuously for 10 days within 12 weeks prior to the study enrollment
* Prior and concomitant immunosuppressants treatment (other than glucocorticoids)
* History and current serious psychiatric disorders that could affect treatment adherence
* Co-existing uncontrolled cardiovascular disease (i.e arterial hypertension), respiratory insufficiency, acute or chronic renal failure (creatinine clearance < 60 ml/min), and liver diseases such as acute or chronic viral hepatitis, alcoholic liver disease, choledocholithiasis, autoimmune hepatitis, non-alcoholic fatty liver disease, hemochromatosis, and liver failure.
* Known history of cholecystitis
* Pregnant or lactating women
* Known hypersensitivity to UDCA, or other bile acids
* History of malignancy diagnosed or treated within 2 years (recent localized treatment of squamous or non-invasive basal skin cancers is permitted; cervical carcinoma in situ is allowed if appropriately treated prior to Screening)
* Participation in any other interventional study

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Change in oxidative stress biomarkers levels: superoxide dismutase (SOD), catalase, and malondialdehyde (MDA) | From Baseline and after 8 weeks
  ELISA assay (same units)
Change in pro-inflammatory markers concentrations: tumor necrosis factor-α (TNF-α), and interleukin 6 (IL-6) | From Baseline and after 8 weeks
  ELISA assay (same units)
Change in serum levels of homocystein | From Baseline and after 8 weeks
  Detection by fluorescence polarization immunoassay
Change in serum levels of von Willebrand factor (vWF), Intercellular Adhesion Molecule 1 (ICAM-1), Vascular Adhesion Molecule 1 (VCAM-1), and fibrinogen | From Baseline and after 8 weeks
  ELISA assay (same units)
Change in serum levels of Vitamin D and Folic acid | From Baseline and after 8 weeks
  Microparticle enzyme immunoassay (same units)
Change in Total antioxidant capacity (TAC) level | From Baseline and after 8 weeks
  Results expressed in units μg/ml Trolox equivalents
Change in inflammation marker level: high sensitivity CRP | From Baseline and after 8 weeks
  Turbid metric test

SECONDARY OUTCOMES:
Change in Haemoglobin A1C (HbA1C) | From Baseline and after 8 weeks
  HbA1C level will be expressed in %
Change in Total cholesterol (TC), low-density lipoprotein (LDL), high-density lipoprotein (HDL), and triglycerides | From Baseline and after 8 weeks
  Clinical biochemistry (colorimetric) tests, and results will be expressed in mmol/L (same units)
Change in body weight | From Baseline and after 8 weeks
  Weight (kg)

CONTACTS AND LOCATIONS:
Overall Officials: Ranko Skrbic, Professor, Study Chair — University of Banja Luka
Locations (1):
- Public Health Institution Dom zdravlja Banja Luka, Banja Luka, Republika Srpska, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lakic B, Skrbic R, Uletilovic S, Mandic-Kovacevic N, Grabez M, Saric MP, Stojiljkovic MP, Soldatovic I, Janjetovic Z, Stokanovic A, Stojakovic N, Mikov M. Beneficial Effects of Ursodeoxycholic Acid on Metabolic Parameters and Oxidative Stress in Patients with Type 2 Diabetes Mellitus: A Randomized Double-Blind, Placebo-Controlled Clinical Study. J Diabetes Res. 2024 Feb 29;2024:4187796. doi: 10.1155/2024/4187796. eCollection 2024. PMID 38455850
- See also: Bile acids signaling pathways have become attractive targets for the treatment of various metabolic diseases and metabolic syndrome opening the new potential avenue in their treatment. — https://pubmed.ncbi.nlm.nih.gov/30559664/